CLINICAL TRIAL: NCT01299675
Title: SureScan Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: SureScan PAS
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Bradycardia
Keywords: MR conditional
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Performance: Subjects enrolled prior to or within 30 days post implant of SureScan pacing system. In office follow-up visits required every 6 months.
- Multiple MRI Scan Characterization: Subject enrolled into study at the time of MRI Scan indication. Subject followed per clinic standard of care.

SUMMARY:
The purpose of this Post-Approval Study (PAS) is to demonstrate the chronic performance of the SureScan pacing system when used in an MRI environment according to product labeling. This study is required by the Food and Drug Administration (FDA) as a condition of product approval.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
2. Subject is or intended to be implanted with a complete SureScan pacing system consisting of both a right atrial and ventricular 5086MRI Lead (used for pacing and sensing) and a SureScan device
3. Subject within 30 days of implant (maximum 50% of Chronic Performance Arm enrollment) or subject enrolled into Multiple MRI Scan Arm at the time of MRI scan indication

Exclusion Criteria:

1. Subject who is, or will be inaccessible for follow-up
2. Implant and follow-up data, including adverse device effects and system modifications at implant through the time of enrollment are unavailable
3. Subject with exclusion criteria required by local law

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients indicated for or implanted with a Medtronic SureScan Pacing System. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2483 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
MRI Related Complication Rate | 5 years
Lead Related Complication Rate | 5 years

SECONDARY OUTCOMES:
Assess change in pacing thresholds after multiple MRI scans | 5 years
Summarize MRI system and scan conditions | 5 years
Pacing system related events | 5 years
Characterize lead impedance | 5 years

CONTACTS AND LOCATIONS:
Locations (61):
- United States (59):
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - East Palo Alto, California
  - Fresno, California
  - Glendale, California
  - Long Beach, California
  - Los Angeles, California
  - Salinas, California
  - Santa Rosa, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - New Haven, Connecticut
  - Bradenton, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Atlanta, Georgia
  - Urbana, Illinois
  - Evansville, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Salisbury, Maryland
  - Takoma Park, Maryland
  - Marquette, Michigan
  - Troy, Michigan
  - Coon Rapids, Minnesota
  - Robbinsdale, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Henderson, Nevada
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Huntington, New York
  - New York, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Elyria, Ohio
  - Toledo, Ohio
  - Bethlehem, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Wyomissing, Pennsylvania
  - Florence, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Milwaukee, Wisconsin
- Canada (2):
  - Kingston, Ontario
  - Trois-Rivières, Quebec

REFERENCES:
- [Derived] Williamson BD, Gohn DC, Ramza BM, Singh B, Zhong Y, Li S, Shanahan L; SureScan Post-Approval Study Investigators. Real-World Evaluation of Magnetic Resonance Imaging in Patients With a Magnetic Resonance Imaging Conditional Pacemaker System: Results of 4-Year Prospective Follow-Up in 2,629 Patients. JACC Clin Electrophysiol. 2017 Nov;3(11):1231-1239. doi: 10.1016/j.jacep.2017.05.011. Epub 2017 Sep 13. PMID 29759618